CLINICAL TRIAL: NCT05544643
Title: Safety and Efficacy of Medtronic Extended Mio 30 Infusion Set
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Prof. Amir Tirosh, Prof. Amir Tirosh, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Sheba-21-8739-at-ctil
Record Dates: First submitted 2022-09-08; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - M30IS vs. EM30IS. First phase Mio 30, second phase Extended Mio 30. (Experimental): Subjects will be randomized to a group who will be using the Mio 30 infusion set (M30IS) for the Phase 1. All patients will be retrained on the use of the M30IS by site staff and will be asked to demonstrate proficiency. All subjects will be instructed to change sets every 3 days or at set failure (replace with another M30IS).
  At day 12 or after using 4 sets (set used defined as a set that was used for more than 6 hours), the patients will return to a visit, return all the extracted catheters sets and will switch to the Extended Mio 30 infusion set (EM30IS), entering Phase 2. All patients will be trained at this visit on the use of the EM30IS by site staff and demonstrate proficiency in the use of the EM30IS. All subjects will be instructed to change sets every 7 days or at set failure (replace with another EM30IS). After 28 days or after using 4 sets, the patients will return all the extracted catheters sets.
  Interventions: Device: Medtronic Extended Mio 30 Infusion Set
- B - EM30IS vs. M30IS. First phase Extended Mio 30, second phase Mio 30 (Experimental): Subjects will be randomized to a group who will be using the EM30IS for the initial Phase. All patients will be trained on the use of the EM30IS by site staff and will be asked to demonstrate proficiency. All subjects will be instructed to change sets every 7 days or at set failure (replace with another EM30IS).
  At day 28 or after using 4 sets (set used defined as a set that was used for more than 6 hours), the patients will return to a visit, return all the extracted catheters sets and will switch to the M30IS, entering Phase 2. All patients will then be retrained on the use of the M30IS by site staff and demonstrate proficiency. All subjects will be instructed to change sets every 3 days or at set failure (replace with another M30IS). After 12 days or after using 4 sets, the patients will all the extracted catheters sets.
  Interventions: Device: Medtronic Extended Mio 30 Infusion Set

INTERVENTIONS:
Device: Medtronic Extended Mio 30 Infusion Set — Safety and Efficacy of Medtronic Extended Mio 30 Infusion Set
  Other Names: Medtronic Mio 30 Infusion Set; Medtronic Quick set infusion set

SUMMARY:
The purpose of this study is to evaluate the Extended Mio 30 infusion set (EM30IS) 7-day functioning compared to the regular Mio 30 infusion set (M30IS) 3-day functioning. The study will be carried out in adult patients with type 1 diabetes.

Secondary objective, to evaluate the differences in glucose control between the infusion set currently used by participants (Medtronic Quick set infusion sets) and the Medtronic Mio 30 Infusion Set.

DETAILED DESCRIPTION:
This is a 1-center, prospective, open-label, cross-over controlled study with type 1 patients with diabetes on insulin pump therapy with Continuous Glucose Monitoring (CGM).

A total of up to 40 subjects will be enrolled in order to have 20 subjects meeting eligibility criteria. Eligible patients meeting the enrollment and randomization criteria will enter a run-in period of up to 1 month for device adaptation. After the run- in phase, The participants will enter the first study part; participants will be randomized into 2 arms, each arm will undergo 2 phases. In each phase a different type of infusion set will be evaluated. Each evaluation will be for 1 month. The order will be determined by the randomization process:

Arm A: Quick set infusion set- M30IS. First phase Quick set, second phase Mio 30.

Arm B: M30IS- Quick set infusion set. First phase Mio 30, second phase Quick set infusion set.

Trial Arm A: Subjects will be randomized to a group who will be using the Quick set infusion set for the initial Phase. All patients will be trained on the use of the Quick set infusion set by site staff and will be asked to demonstrate proficiency. All subjects will be instructed to change sets every 3 days or at set failure (replace with another Quick set infusion set).

After 1 month, the patients will return to a visit, return all the extracted catheters sets and will switch to the M30IS, entering Phase 2. All patients will then be retrained on the use of the M30IS by site staff and demonstrate proficiency. All subjects will be instructed to change sets every 3 days or at set failure (replace with another M30IS). 1 month, the patients will return all the extracted catheters sets.

Trial Arm B: Subjects will be randomized to a group who will be using the Mio 30 infusion set (M30IS) for the second Phase. All patients will be retrained on the use of the M30IS by site staff and will be asked to demonstrate proficiency. All subjects will be instructed to change sets every 3 days or at set failure (replace with another M30IS).

After 1 month, the patients will return to a visit, return all the extracted catheters sets and will switch to the Quick set infusion set, entering Phase 2. All patients will be trained at this visit on the use of the Quick set infusion set by site staff and demonstrate proficiency in the use of the Quick set infusion set. All subjects will be instructed to change sets every 3 days or at set failure (replace with another Quick set infusion set). 1 month, the patients will return all the extracted catheters sets

After completing the first study part, participants will be randomized again into 2 arms, each arm will undergo 2 phases. In each phase a different type of infusion set will be evaluated. Each evaluation will be for 4 sets (up to 28 days). The order will be determined by the randomization process:

* Arm A: M30IS - EM30IS. First phase Mio 30, second phase Extended Mio 30.
* Arm B: EM30IS - M30IS. First phase Extended Mio 30, second phase Mio 30. Trial Arm A: Subjects will be randomized to a group who will be using the Mio 30 infusion set (M30IS) for the Phase 1. All patients will be retrained on the use of the M30IS by site staff and will be asked to demonstrate proficiency. All subjects will be instructed to change sets every 3 days or at set failure (replace with another M30IS).

At day 12 or after using 4 sets (set used defined as a set that was used for more than 6 hours), the patients will return to a visit, return all the extracted catheters sets and will switch to the Extended Mio 30 infusion set (EM30IS), entering Phase 2. All patients will be trained at this visit on the use of the EM30IS by site staff and demonstrate proficiency in the use of the EM30IS. All subjects will be instructed to change sets every 7 days or at set failure (replace with another EM30IS). After 28 days or after using 4 sets, the patients will return all the extracted catheters sets.

Trial Arm B: Subjects will be randomized to a group who will be using the EM30IS for the initial Phase. All patients will be trained on the use of the EM30IS by site staff and will be asked to demonstrate proficiency. All subjects will be instructed to change sets every 7 days or at set failure (replace with another EM30IS).

At day 28 or after using 4 sets (set used defined as a set that was used for more than 6 hours), the patients will return to a visit, return all the extracted catheters sets and will switch to the M30IS, entering Phase 2. All patients will then be retrained on the use of the M30IS by site staff and demonstrate proficiency. All subjects will be instructed to change sets every 3 days or at set failure (replace with another M30IS). After 12 days or after using 4 sets, the patients will all the extracted catheters sets.

Each subject will wear MiniMed™ 780G/670G insulin system. Each subject will be given for the first study part: 11 infusion sets each to wear, each infusion set for at least the labelled use time (3 days for M30IS or 3 days for Quick set infusin set), or until infusion set failure if this occurs before 3 days.for the second part 4 infusion sets each to wear, each infusion set for at least the labelled use time (3 days for M30IS or 7 days for EM30IS), or until infusion set failure if this occurs before 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least one year
* Age 18 to 80 years
* Not currently known to be pregnant, nor planning pregnancy during the study.
* Willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.
* Pregnant or lactating females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Percentage of sets that failed due to unexplained hyperglycemia | 6 months
  The primary outcome is to have no more than 16% of infusion set failures due to "unexplained hyperglycemia"

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Sheba Medical Center, Ramat Gan
  - Sheba Medical Center, Tel Litwinsky